CLINICAL TRIAL: NCT04171778
Title: Effects of a Whole Food, Plant-Based Nutrition Program on Subjects With Chronic Kidney Disease and Proteinuria
Brief Title: Effects of Whole Food, Plant-Based Nutrition on Chronic Kidney Disease With Proteinuria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Substantially redesigning study protocol and opening a new study in the future.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Erin Campbell, Clinical Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003490
Record Dates: First submitted 2019-10-29; First posted 2019-11-21 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease Stage 3B; Chronic Kidney Disease, Stage 4; Proteinuria
Keywords: CKD; proteinuria; diet; plant-based diet; vegan; randomized controlled trial
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: The initial phase of the study will be a three month randomized clinical trial of a whole food plant based nutrition program vs. usual care in patients with chronic kidney disease. Subjects randomized to the intervention arm will start the nutrition program as soon as they are able.
  Subjects assigned to the control arm will be placed on a 'wait-list' to start the nutrition program after they undergo three months of testing during their usual care, which consists of routine CKD care as directed by their primary nephrologist. After a 3 month 'wait', they will start the same plant-based nutrition program as the intervention arm subjects.
  Both experimental and control group subjects will be followed for a total of 9 months after starting the plant-based dietary intervention. Thus, in addition to the 3-month randomized control trial, there will be data from a 9-month single arm clinical intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects in this arm will immediately begin a whole-food, plant-based nutrition program consisting of weekly educational group meetings and prepared meals delivered to the subjects' homes for the first 12 weeks followed by monthly educational group meetings for an additional 6 months.
  Interventions: Other: whole food, plant-based diet
- Wait List Control (Other): Subjects in this arm will continue their usual care as directed by their nephrologist for 12 weeks before starting the same whole-food, plant-based nutrition program as the intervention arm subjects.
  Interventions: Other: whole food, plant-based diet

INTERVENTIONS:
Other: whole food, plant-based diet — The study diet is whole food, plant based defined as containing no animal products or refined grains or added oils, minimal use of any sweeteners, and, for the purposes of this study, on average containing no more than 15% calories from fat.

SUMMARY:
This study will test the hypothesis that lifestyle intervention consisting of a whole food, plant-based (WFPB) diet and group education will favorably impact outcomes germane to individuals with chronic kidney disease (CKD) stage 3b and 4, including blood pressure control, amount of proteinuria (protein in the urine), and preservation of glomerular filtration rate (GFR). In addition, this study will assess weight and body composition, diabetic control in subjects with diabetes as well as CKD, and quality of life. Safety of a WFPB diet in subjects with CKD will be tested with respect to the development of elevated serum potassium and phosphorus, hypoalbuminemia (low blood protein), hypotension (low blood pressure), and hypoglycemia (low blood sugar). An exploratory aim is to test the effects of a WFPB diet on the microbiome of subjects by collecting and analyzing stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Subjects with CKD 3b and 4 (as determined by an estimated glomerular filtration rate of ≥ 15 ml/min but ≤ 45 ml/min for at least three months)
* Subjects with proteinuria documented at least twice with the most recent test within the last 6 months as determined by:

  * Urine albumin excretion rate of > 300 mg/day or urine albumin to creatinine ratio of > 300 mg/g of creatinine
  * Urine protein excretion rate of > 500 mg/day or urine protein to creatinine ratio of > 0.5 g/g of creatinine
* If using angiotensin converting enzyme inhibitor, angiotensin receptor blockers and/or aldosterone antagonists, on a stable dose of for greater than one month
* Fluent in English language
* Able and willing to comply with the testing and group education schedules
* Able and willing to comply with a whole-food, plant-based diet
* Able and willing to give informed consent

Exclusion Criteria:

* Any kidney disease requiring immunosuppressive therapy
* Pregnancy or intent to become pregnant in the next 12 months
* Life expectancy < 12 months
* History of solid organ transplant or anticipated solid organ transplant in next 12 months
* History of hyperkalemia: Two potassium measurements > 5.1 Meq/L within the last three months, or history of any intervention for hyperkalemia in the last 6 months
* Subjects with malabsorptive syndromes
* Subjects with history of bariatric surgery or planned bariatric surgery in the next 12 months
* Subjects on warfarin
* Subjects with current eating disorders
* Subjects with tobacco or illicit substance use
* Subjects with alcohol use of > 7 drinks per week
* Allergy or intolerance of a plant-based or plant-derived food (gluten, soy, etc.)
* Following a vegan diet in the six months prior to consent
* Major surgery within 60 days prior to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure from baseline | 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Change in proteinuria from baseline | 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Urine total protein:creatinine ratio
Change in GFR from baseline | 1, 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Serum creatinine (renal function panel) and Cystatin C

SECONDARY OUTCOMES:
Weight changes from baseline | 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
BMI changes from baseline | 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Waist circumference changes from baseline | 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
8-point bioelectrical impedance analysis changes from baseline | 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Body composition assessment
Hemoglobin A1c changes from baseline | 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Diabetic control
KDQOL-36 changes from baseline | 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Scoring of this questionnaire consists of 5 scales (symptoms/problem list, effects of kidney disease, burden of kidney disease, SF-12 physical composite, and SF-12 mental composite). The lowest possible score for each scale is 0, indicating the worst outcome, and the best possible score is 100, indicating the best possible outcome.
Serum potassium changes from baseline | 1, 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Serum phosphorus changes from baseline | 1, 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Serum albumin changes from baseline | 1, 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Blood glucose level changes from baseline | 1, 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Fasting serum levels from all subjects; additionally, whole blood levels measured by glucometer in subjects with comorbid type 1 or type 2 diabetes mellitus
Total cholesterol, HDL, LDL, and non-HDL cholesterol level changes from baseline | 1, 4, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Fasting lipid panel
Serum magnesium changes from baseline | 1, 4, 8, and 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Parathyroid hormone (PTH) changes from baseline | 12 weeks (RCT); 3 and 9 months on intervention diet (all subjects)
25-hydroxycholecalciferol changes from baseline | 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Fibroblast growth factor-23 changes from baseline | 12 weeks (RCT); 3 and 9 months on intervention diet (all subjects)
High sensitivity CRP changes from baseline | 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
CBC with differential changes from baseline | 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
Changes in nutrient intakes from baseline based on 3 day food diaries | 12 weeks (RCT); 3, 6, and 9 months on intervention diet (all subjects)
  Assess baseline compared to intervention diet and assess compliance of intervention diet over study duration
Changes in urinary indicators of dietary intake from baseline | 12 weeks (RCT); 3 and 9 months on intervention diet (all subjects)
  24 hour urine collection, urinary oxidation (urinary 8-isoprostane)

OTHER OUTCOMES:
Exploratory stool microbiome evaluation | 12 weeks (RCT)
  Changes in microbiome from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Erin Campbell, MD, MPH, Principal Investigator — University of Rochester; Scott E Liebman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Highland Hospital (University of Rochester), Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available for collaboration or other purposes with appropriate data use agreements in place.